CLINICAL TRIAL: NCT00506597
Title: Erwinia L-Asparaginase (Erwinase) Study in Patients With Acute Lymphoblastic Leukemia
Brief Title: Erwinase Study in Patients With Acute Lymphoblastic Leukemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0183
Record Dates: First submitted 2007-07-20; First posted 2007-07-25 (Estimated); Results first posted 2014-09-11 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Leukemia
Keywords: Acute Lymphoblastic Leukemia; Leukemia; Erwinia L-Asparaginase; Erwinase
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Asparaginase; asparaginase erwinia chrysanthemi recombinant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Erwinase (Experimental): 6 doses of 25,000 Units/m^2 Erwinase® intramuscular/subcutaneously every other day to replace each dose of Pegylated Asparaginase
  Interventions: Drug: Erwinase

INTERVENTIONS:
Drug: Erwinase — If allergic to E.Coli Asparaginase = 1 Dose (20,000 Units/m^2) Daily; If allergic to Pegylated Asparaginase = 6 Doses (25,000 Units/m^2) Daily Every Other Day. Received as an injection through a needle in vein, under the skin, or in muscle.
  Other Names: Erwinia L-Asparaginase

SUMMARY:
The goal of this clinical research study is to allow doctors to use Erwinia L-Asparaginase (Erwinase®) as a replacement for patients who are allergic to E.coli L-asparaginase or Pegylated E.coli L-asparaginase as part of the treatment for acute lymphoblastic leukemia (ALL) or T or B cell lymphoma.

This trial was part of a multi institutional effort by the drug company to make Erwinase available for use.

DETAILED DESCRIPTION:
The Study Drug:

Erwinia L-Asparaginase helps stop the growth of cancer cells by blocking the nutrients that cancer cells needed to survive.

Study Visits:

Erwinia L-Asparaginase will be given either outpatient or inpatient, depending upon your condition.

If you are allergic to E. Coli Asparaginase or Pegylated Asparaginase, you will be given 6 doses every other day.

You will receive Erwinia L-Asparaginase as an injection through a needle in your vein, under the skin, or in your muscle, as directed by your study doctor.

You will be monitored closely by your nurse and your doctor before, during, and after receiving the drug for any side effects. If you develop a severe allergy to Erwinia L-Asparaginase, you may not receive any more asparaginase therapy.

The length of study will be based upon on the ALL treatment you are currently receiving. Your doctor will discuss the details of your treatment schedule with you.

This is an investigational study. Erwinia L-Asparaginase is not FDA approved. The FDA allows patients with acute lymphoblastic leukemia who have an allergic reaction to the U.S.-approved L-asparaginases to receive Erwinia L-Asparaginase. Up to 35 patients will take part in this study at The University of Texas (UT) MD Anderson Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

1. Age: no restrictions
2. Patient must give written informed consent to receive Erwinase® under Investigational New Drug (IND) 290.
3. Patient must be treated for Acute Lymphoblastic Leukemia
4. Patient with either T or B cell lymphoma being treated with Asparaginase.
5. Patient must have either systemic hypersensitivity reactions to native (Elspar®) or pegylated (Oncaspar®) E. coli L-Asparaginase. This includes patients with generalized rash with or without anaphylactic symptoms, but not those with only local pain or redness at the site of injection.
6. Patient with previously documented local or systemic reactions to E. coli derived L-Asparaginase.
7. Patients who are on Elspar® (including those enrolled in a clinical trial randomized to Elspar®) and where Elspar® is not available.

Exclusion Criteria:

1. Previous allergic reaction to Erwinia L-Asparaginase (Erwinase ®)
2. Previous acute pancreatitis
3. Pregnant or lactating woman

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2007-05; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J. Wells, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas MD Anderson Cancer Center Official Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The University of Texas (UT) MD Anderson Cancer Center Recruitment Period: May 07, 2007 to November 29, 2011. Recruitment site specifically at MD Anderson Cancer Center medical clinics.
Pre-assignment Details: This trial was part of a multi institutional effort by the drug company to make Erwinase available for use. The participants reported were recruited and treated as part of the trial site participation at MD Anderson Cancer Center.
Period: Overall Study
Arm/Group | Erwinase
Started | 33
Completed | 33
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Erwinase
Number analyzed (Participants) | 33
Age, Continuous [Median (Full Range); unit: years] | 15 [2 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 19
Region of Enrollment [Number; unit: participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Participant Toxicity Data
Description: Toxicity data collected and reported as adverse events during the study period. See Adverse Event section for reporting.
Time Frame: 3 Years
Reporting Status: Not Posted

2. Primary Outcome: Number of Participants Treated With Erwinase as a Replacement for E.Coli L-asparaginase or Pegylated E.Coli L-asparaginase as Part of the Treatment for Acute Lymphoblastic Leukemia (ALL) or T or B Cell Lymphoma
Description: Main objective of protocol Erwinase® Master Treatment Protocol (EMTP) was to enable United States (US) participants who were treated for Acute Lymphoblastic Leukemia (ALL) and who were allergic to Escherichia coli derived L-Asparaginase, whatever the formulation, to be treated with Erwinia derived L-Asparaginase (Erwinase®), under Investigational New Drug (IND) 290.
Time Frame: 4 years
Measure: Number; unit: participants
Arm/Group | Erwinase
Number analyzed (Participants) | 33
participants | 33

ADVERSE EVENTS:
Time Frame: Adverse event data collected during administration of 6 doses of Erwinase® intramuscular/subcutaneously every other day to replace each dose of Pegylated Asparaginase. Overall study period 3 years and 5 months.
Arm/Group | Erwinase
Serious Adverse Events (participants affected / at risk) | 7/33
Other Adverse Events (participants affected / at risk) | 6/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erwinase (N=33)
Hyperglycemia (Blood and lymphatic system disorders) | 1
White Blood Count Decreased (Blood and lymphatic system disorders) | 1
Cardiopulmonary Failure (Cardiac disorders) | 1
Infection (Infections and infestations) | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erwinase (N=33)
Allergic Reaction (Immune system disorders) | 1
Fever/Infection (Infections and infestations) | 1
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1
Parathesia (Musculoskeletal and connective tissue disorders) | 1
Facial Weakness (Musculoskeletal and connective tissue disorders) | 1
Headache (General disorders) | 1
Prothrombin time (PTT) increased (Blood and lymphatic system disorders) | 1
Pancreatitis (Endocrine disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No